CLINICAL TRIAL: NCT06261281
Title: A Randomized Controlled Study to Explore the Effect of Intermittent Oro-esophageal Tube Feeding on Severe Traumatic Brain Injury Patient
Brief Title: Effect of Intermittent Oro-esophageal Tube Feeding on Severe Traumatic Brain Injury Patient
Acronym: IOE-TBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical issue
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBI cancel
Record Dates: First submitted 2024-01-28; First posted 2024-02-15 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The observation group (Experimental): Both groups of patients were provided with routine treatments, including pharmacological treatment, rehabilitation therapy.Based on this, the patients in the observation group were given enteral nutrition support with Intermittent Oro-esophageal Tube Feeding (Medical Device No. 20010234, developed by the Swallowing Disorders Research Institute of Zhengzhou University).
  Interventions: Behavioral: Rehabilitation therapy; Device: Intermittent Oro-esophageal Tube Feeding
- The control group (Active Comparator): Both groups of patients were provided with routine treatments, including pharmacological treatment, rehabilitation therapy. The patients in the control group were provided nutrition support with Nasogastric tube feeding , while the feeding process strictly followed the relevant guideline
  Interventions: Behavioral: Rehabilitation therapy; Device: Nasogastric tube feeding

INTERVENTIONS:
Behavioral: Rehabilitation therapy — Including:Acupuncture: Regular acupuncture treatment that can prevent muscle atrophy, improve circulation, and have a stimulating effect. Exercise therapy: Training that focused on limb movements or joint mobilization to prevent muscle contracture, reduce joint mobility, improve spasms, and promote blood circulation. Others: Regular turning, back patting, and position changes performed by caregivers.
Device: Intermittent Oro-esophageal Tube Feeding — Based on this, the patients in the observation group were given nutrition support with Intermittent Oro-esophageal Tube Feeding (Medical Device No. 20010234, developed by the Swallowing Disorders Research Institute of Zhengzhou University). The entire feeding process strictly followed the standard procedure of Intermittent Oro-esophageal Tube Feeding. During the feeding process, patients were maintained in a semi-recumbent position with their head elevated, facilitating the placement of the tube into the oral cavity along one side, with the chin brought close to the manubrium sterni.
  Arms: The observation group
Device: Nasogastric tube feeding — The patients in the control group were provided nutrition support with Nasogastric tube feeding, while the feeding process strictly followed the relevant guideline. During the treatment, the patients remained in a continuous state of tube indwelling, receiving feeding every 2-3 hours with a maximum feeding volume of 200ml, of which the contents were consistent with the observation group. The entire feeding process was conducted by trained nursing staff. Besides, the tube was replaced by a new one every 5-7 days.
  Arms: The control group

SUMMARY:
This was a multicenter randomized controlled study of 98 severe Traumatic Brain Injury patients with tracheostomy. Patients enrolled were divided randomly into the observation group with Intermittent Oro-esophageal Tube Feeding or the control group with Nasogastric tube feeding for enteral nutrition support, respectively. Nutritional status, complications, decannulation of tracheostomy tubes and level of consciousness on day 1 and day 28 were recorded and compared.

DETAILED DESCRIPTION:
The safe and effective nutrition support for severe traumatic brain injury patients with tracheostomy continues to be a challenge. Nasogastric tube feeding has been the mainstream choice in China but with the risk of complications. Intermittent Oro-esophageal Tube Feeding is an established modality of enteral nutrition support that can be used with routine treatment. This study reports the clinical outcomes of Intermittent Oro-esophageal Tube Feeding vs. nasogastric tube feeding, in patients receiving routine treatment. This was a multicenter randomized controlled study of 98 severe traumatic brain injury patients with tracheostomy. Patients enrolled were divided randomly into the observation group with Intermittent Oro-esophageal Tube Feeding or the control group with Nasogastric tube feeding for enteral nutrition support, respectively. Nutritional status, complications, decannulation of tracheostomy tubes and level of consciousness on day 1 and day 28 were recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years, meeting the diagnosis of severe Traumatic Brain Injury, confirmed through MRI
* score of Glasgow Coma Scale (GCS) <8;
* presence of no contraindication for enteral nutrition;
* with stable vital signs and no severe liver or kidney dysfunction, metabolic disorders, cardiovascular diseases, or multiple complications;
* informed consent form was obtained from the patients' family members, indicating their full understanding of the study and agreement to participate.

Exclusion Criteria:

* unable to cooperate in completing treatment and assessment due to personal reasons or other disorders;
* complicated with other intracranial lesions, such as stroke;
* with severe consciousness disorders caused by other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Concentration of hemoglobin | day 1 and day 28
  hemoglobin was tested with blood routine test
Concentration of albumin | day 1 and day 28
  albumin was tested with blood routine test
Concentration of prealbumin | day 1 and day 28
  prealbumin was tested with blood routine test
Nutritional status-body mass index | day 1 and day 28
  body mass index was tested with body weight and height. Combination was calculated as: body weight (kg) / height (m)^2.

SECONDARY OUTCOMES:
Decannulation of tracheostomy tube-placement duration | day 1 and day 28
  The duration of tracheostomy tube retention and the outcomes of decannulation were recorded for two groups during the treatment. The criteria for tracheostomy tube removal were as follows: patients should exhibit no significant pulmonary complications (including the progressive decline in blood oxygen, carbon dioxide retention, pneumonia, etc.) during the capping trial, and should exhibit stable, regular breath and not require reintubation or tracheostomy within 72 hours after tube removal.
Decannulation of tracheostomy tube-Successful removal | day 1 and day 28
  The duration of tracheostomy tube retention and the outcomes of decannulation were recorded for two groups during the treatment. The criteria for tracheostomy tube removal were as follows: patients should exhibit no significant pulmonary complications (including the progressive decline in blood oxygen, carbon dioxide retention, pneumonia, etc.) during the capping trial, and should exhibit stable, regular breath and not require reintubation or tracheostomy within 72 hours after tube removal
Level of consciousness | day 1 and day 28
  The Glasgow Coma Scale was used to assess the level of consciousness in patients. A score of 15 indicates normal consciousness, a score of 13-14 indicates mild consciousness impairment, a score of 9-12 indicates moderate consciousness impairment, and a score less than 8 indicates severe consciousness impairment.
Feeding Amount | day 1 and day 28
  The total amount of nutrients consumed by the patient on the day was recorded, excluding fresh water, units: milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Tian, Doctor, Study Chair — Zhengzhou University
Locations (1):
- Zheng Da yi Yuan Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No